CLINICAL TRIAL: NCT05209724
Title: Remote Monitoring of Home Exercise in Peripheral Arterial Disease
Acronym: ROMEPAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dallas VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Subhash Banerjee, Principal Investigator, Dallas VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1602740
Record Dates: First submitted 2022-01-13; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Peripheral Arterial Disease
Keywords: PAD; Home walking; Remote monitoring; Claudication
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Provider Supervised (Experimental): Digital monitoring system with provider supervision
  Interventions: Behavioral: Provider supervision/ feedback
- Self Supervised (No Intervention): Digital monitoring system without provider supervision

INTERVENTIONS:
Behavioral: Provider supervision/ feedback — Provider supervision/ feedback provided before and after walking sessions
  Arms: Provider Supervised

SUMMARY:
Many patients with blockages in the arteries in their legs (peripheral arterial disease, "PAD") suffer from pain in their legs when walking. Exercise therapy is known to decrease pain levels as well as increase the distance that patients with PAD can walk. The purpose of this study is to understand whether home exercise using a digital exercise monitoring system (LIVMOR) with provider supervision/ feedback will improve walking distance compared to those undergoing home exercise using the same monitoring system but without provider supervision/ feedback.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Diagnosis of PAD (based on ABI <0.9 in either leg or prior intervention) with mild/moderate claudication

Exclusion Criteria:

* Prior above ankle amputation
* Wheelchair bound
* Inability to walk >200m during 6 min walk test
* Use of walking aid other than cane
* Walking impairment for reason other than PAD
* Critical limb ischemia
* Planned vascular surgery within next 3 months, recent surgery within past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2021-11-21 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Change in 6 minute walk test distance between groups | 12 weeks
  Change in 6 minute walk test distance between groups

SECONDARY OUTCOMES:
Change in Walking Impairment Questionnaire score | 12 weeks
  Change in Walking Impairment Questionnaire score between groups
Change in VascuQOL-6 (VQ6) quality of life survey | 12 weeks
  Change in VascuQOL-6 (VQ6) quality of life survey between groups

CONTACTS AND LOCATIONS:
Overall Officials: Subhash Banerjee, MD, MBA, Principal Investigator — Dallas VA Hospital
Locations (1):
- Dallas North Texas Veterans Affairs Hospital, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No IPD are to be shared.